CLINICAL TRIAL: NCT02292602
Title: Developing a Preschool Obesity Intervention for Families Enrolled in WIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: Michigan Department of Community Health (Other)
Responsible Party: Principal Investigator, Elizabeth Kuhl, Assistant Professor of Pediatrics, Wayne State University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21HD078890-01 (NIH)
Record Dates: First submitted 2014-11-09; First posted 2014-11-17 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Pediatric Obesity
Keywords: preschool; obesity; health disparities; intervention
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family-Based Weight Control Intervention (Experimental): Families will receive the FBWC
  Interventions: Behavioral: Family-Based Weight Control
- Control (No Intervention): Families will continue with standard of care at WIC

INTERVENTIONS:
Behavioral: Family-Based Weight Control — Families randomized to the intervention condition will receive a 4-month, 14-session behavioral weight control intervention targeting obesity reduction in preschoolers and caregivers. Within the program, 9 sessions will be group-based and held at WIC and 5 sessions will be individual visits (4 home-based and 1 at a food market where the family shops). The intervention includes teaching behavioral weight loss, child behavior management, and life skills (e.g., budgeting and time management ) via experiential learning to assist families with implementing diet and activity recommendations for pediatric and adult weight management.
  Other Names: FBWC
  Arms: Family-Based Weight Control Intervention

SUMMARY:
The purpose of this study is to examine the feasibility, acceptability, and preliminary efficacy of a community and home-based preschool obesity intervention for families enrolled in the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC).

DETAILED DESCRIPTION:
Very few studies have targeted weight control in preschoolers even though the prevalence of overweight has exceeded 20% in this age-group for the past decade. Also concerning is that few studies have focused on preschoolers from low-socioeconomic (SES) backgrounds despite persistent obesity-related socioeconomic disparities. Family-based, behavioral interventions appear a promising model for treatment of obesity in early childhood. However, the dissemination potential of these programs is unclear as they have primarily been tested with families from middle-to-upper class backgrounds and within research settings. Identifying effective approaches to weight control for preschoolers from low-SES backgrounds that can be delivered in community settings is imperative to reducing the pediatric obesity epidemic. The proposed study will begin to address this critical gap by completing the second phase of developing a community-based preschool weight control intervention for families enrolled in the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC). The proposed study is significant because we specifically target preschool weight control in a high-risk population and because delivery of our program within the WIC program is conducive to its dissemination. Based upon our formative work, and existing preschool obesity programs, we have developed a 14-session, family-based preschool weight control intervention (FBWC) that emphasizes experiential learning and is delivered in the WIC and home settings. Seventy-two overweight and obese preschool-caregiver dyads will be randomized in a 2:1 ratio to receive FBWC or to continue with standard of care at WIC (WSOC). The primary study aims are to a) examine the feasibility and acceptability of FBWC and b) explore the preliminary efficacy of FBWC compared to WSOC on reduction in preschooler BMI-z-score and caregiver BMI from baseline to post-treatment (4-months) and 7-months (3-month follow-up). An exploratory aim is to evaluate lifestyle and behavioral indicators of intervention success. This study is innovative because: 1) very few studies have examined obesity intervention in preschoolers, 2) we target weight control in a high-risk group that has been underrepresented in the preschool obesity treatment outcome literature, 3) our intervention is community-based, and 4) we emphasize experiential learning as a strategy for achieving lifestyle behavior change and weight control.

ELIGIBILITY:
Inclusion Criteria:

* family receiving services at Detroit-based WIC clinics
* preschooler between the ages of 2 years and 4 years, 7 months and BMI>85th percentile
* one primary caregiver who is willing to participate and whose BMI>25
* family is English-speaking
* preschooler has medical clearance to participate in the intervention
* caregiver has medical clearance to participate in the intervention if indicated by physical activity screening questions

Exclusion Criteria:

* preschooler or caregiver is participating in a different weight management program
* preschooler or caregiver has a condition that precludes participation in moderate level activity
* preschooler or caregiver is diagnosed with a weight-affecting health condition
* preschooler or caregiver is taking weight-affecting medications
* preschooler or caregiver is diagnosed with a developmental delay or disability
* caregiver is receiving treatment for severe psychopathology
* family plans to be out of town for more than 2 weeks of the first 4 months of their research participation
* family plans to move from Detroit in the next 7 months

Ages: 24 Months to 55 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2014-02; Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Feasibility (attendance and attrition) | 4-months
  mean number of sessions attended and number of families who dropped out of the intervention
Perceived acceptability of the program at post-treatment as measured by semi-structured qualitative interviews | 4 months
  Semi-structured qualitative interviews will be conducted with a randomly selected subset of families completing the intervention (n=12) to determine whether the intervention met their needs.
Perceived acceptability of the program at follow-up | 7 months
  Semi-structured qualitative interviews will be conducted with a randomly selected subset of families completing the intervention (n=24) to determine whether intervention content facilitated sustained change.
Change in preschooler BMI z-score | baseline, 4 months, 7 months
  based upon height and weight
Change in and caregiver BMI | baseline, 4 months, 7 months
  based upon height and weight

SECONDARY OUTCOMES:
Change in preschooler diet | baseline, 4-months, 7-months
  24-hour dietary recall
Change in preschooler activity | baseline, 4-months, 7-months
  accelerometry
Change in caregiver diet | baseline, 4-months, 7-months
  Block Brief Questionnaire
Change in caregiver activity | baseline, 4-months, 7-months
  Paffenbarger Activity Questionnaire
Change in caregiver feeding | baseline, 4-months, 7-months
  Child Feeding Questionnaire, Caregiver's Feeding Style Questionnaire
Change in caregiver stress | baseline, 4-months, 7-months
  Perceived Stress Scale
Change in home food environment | baseline, 4-months, 7-months
  observational measure of energy- and nutrient-dense foods in the home

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University, Detroit, Michigan, United States